CLINICAL TRIAL: NCT04686513
Title: Relative Risk of Hypertension Among Young Adult Obese Population
Brief Title: Relative Risk of Hypertension Among Obese
Status: Completed | Type: Observational
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Batool Hassan, Principal Investigator, Ziauddin University
Other Study IDs: Batool
Record Dates: First submitted 2020-12-19; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese young adult
  Interventions: Other: Observation
- Non Obese young adult
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — observational study

SUMMARY:
Observational study was conducted to determine the relative risk of hypertension among young adult obese population of Pakistan with age between 25-40 years

ELIGIBILITY:
Inclusion Criteria:

Adult population with age between 25- 40 years having normal weight or Obesity of grade I and II, with or without hypertension.

Exclusion Criteria:

Patients with co-morbid like Diabetes mellitus, dyslipidemia, and cardiovascular disorder were excluded from the study

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese young adult population of BMI <25kg/m2
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Hypertension | day 1
  International Society of Hypertension Global Hypertension Practice Guidelines 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Batool Hassan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No